CLINICAL TRIAL: NCT05267678
Title: A Cohort Study Investigating Nutritional Deficiency Among Pregnant Women With History of Recurrent Miscarriage
Brief Title: Nutritional Deficiency and Recurrent Miscarriage
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Westlake University (Other)
Collaborators: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20220215SHJ001
Record Dates: First submitted 2022-02-21; First posted 2022-03-04 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Recurrent Miscarriage
MeSH Terms: conditions — Abortion, Habitual

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Maternal blood during pregnancy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women with history of recurrent miscarriage
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is an observational study without any intervention

SUMMARY:
This prospective cohort study primarily aims to examine the association between blood niacin levels and recurrent miscarriage.

DETAILED DESCRIPTION:
Recurrent miscarriage is affecting around 5% women at reproductive age. And the underlying causes remain undetermined in 50%-70% of cases. Although animal models and linkage analysis according to family studies have identified that niacin deficiency can lead to congenital malformations and recurrent miscarriage. Evidence based on population is lacking with regard to the effect of blood niacin levels on recurrent miscarriage. We intend to enroll 499 pregnant women confirmed by a positive blood human chorionic gonadotropin test and with history of unexplained recurrent miscarriage. By testing their blood niacin levels and following up to the end of first-trimester pregnancy, this study aims to examine the role of niacin levels in preventing miscarriages among women with history of recurrent miscarriage.

ELIGIBILITY:
Inclusion Criteria:

* 18-40years old, female
* Positive blood human chorionic gonadotropin test
* Naturally pregnant
* History of recurrent miscarriage (2 or more consecutive spontaneous miscarriage within 28 weeks of gestation)
* Willing to participate in this study with informed consent

Exclusion Criteria:

* Women whose confirmed cause of recurrent miscarriage has nothing to do with nutritional deficiencies, including chromosomal abnormalities, abnormal uterine anatomy, immune system diseases, blood diseases, etc.
* Women with Hepatitis B, syphilis, HIV/AIDS and other infectious diseases.
* Women with serious conditions, such as schizophrenia, tumors, heart failure

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women with history of recurrent miscarriage
Sampling Method: Non-Probability Sample
Enrollment: 499 (Estimated)
Dates: Start 2023-01-28 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with miscarriage | 6-13(+6) weeks of gestation
  pregnancy outcomes are confirmed by electronic hospital records or self-reported by participants
Gestation week at miscarriage | 6-13(+6) weeks of gestation
  pregnancy outcomes are confirmed by electronic hospital records or self-reported by participants

CONTACTS AND LOCATIONS:
Overall Officials: Hongjun Shi, PhD, Principal Investigator — Westlake University
Locations (1):
- Peking Union Medical College Hospital, Peking Union Medical College and Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided